CLINICAL TRIAL: NCT00935766
Title: Latinos Using Cardio Health Actions to Reduce Risk (LUCHAR): Effect of Omega-3 Fatty Acids on Vascular Function and Inflammation
Brief Title: Effect of Fish Oil (Omega-3 Fatty Acids) on Arteries
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was discontinued early due to lack of funding and slow enrollment
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Carlin Long, Cardiologist, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-0722 LUCHAR AIM 4
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Diseases; Endocrine System Diseases; Heart Disease; Vascular Diseases; Diabetes; Cardiovascular Disease; Glucose Metabolism Disorders; Hypertension
Keywords: Latinos Using Cardio Health Actions to Reduce Risk; Omega three Fatty Acids; Vascular Function and Inflammation
MeSH Terms: conditions — Metabolic Diseases; Endocrine System Diseases; Heart Diseases; Vascular Diseases; Diabetes Mellitus; Cardiovascular Diseases; Glucose Metabolism Disorders; Hypertension; Inflammation | interventions — Docosahexaenoic Acids; Omacor; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): 4 tabs of placebo dependent on randomization
  Interventions: Drug: Placebo
- Omega 3 (Active Comparator): omega-3-acid ethyl esters and instructed to take 4 1 mg capsules daily
  Interventions: Drug: Omega-3

INTERVENTIONS:
Drug: Omega-3 — Subjects meeting eligibility criteria will be randomized to receive a supply of omega-3-acid ethyl esters or placebo, and instructed to take 4 capsules daily. A 3-month supply of study drug will be given following randomization and at 3, 6, and 9 months. Subjects will be asked to bring unused supplies to each quarterly visit for ascertainment of adherence.
  Other Names: Lovaza
  Arms: Omega 3
Drug: Placebo
  Other Names: Sugar pill
  Arms: Sugar Pill

SUMMARY:
The overall objective of LUCHAR Specific Aims 4.1 and 4.2 is to assess the additional contribution of cardiovascular disease (CVD) risk markers to traditional biomedical risk factors in the prediction of pre-clinical CVD. Specific Aim 4.3 will test the impact of omega-3 fatty acid supplementation on risk markers and pre-clinical markers of CVD in Hispanic patients.

Specific Aim 4.3: Conduct a randomized, placebo-controlled trial of the effect of omega-3 fatty acid supplementation on vascular function as measured by brachial artery reactivity (BAR) and on circulating inflammatory markers.

Hypotheses:

1. Daily omega-3 fatty acid supplementation will improve vascular function in subjects at high risk for CVD.
2. Daily omega-3 fatty acid supplementation will reduce inflammatory protein panel scores in subjects at high risk for CVD.

DETAILED DESCRIPTION:
Omega-3 fatty acids reduce triglycerides (TG) in a manner similar to fibric acids by lowering hepatic TG release, reducing VLDL production, stimulating lipoprotein lipase and enhancing TG clearance. Although statins are widely utilized among DH patients, our overall population, even those with CHD, have fairly low levels of LDL-cholesterol (Krantz et al, 2004). This likely reflects our population that is predominantly Latino with a high incidence of metabolic syndrome. Among our patients, we often achieve LDL-c NCEP targets, yet secondary goals for non-HDL, HDL, and TG are rarely achieved. This is an unmet opportunity given the strong independent contribution of non-HDL (McQueen et al, 2008), HDL (D'Agostino et al, 2008) and TG (Nordestgaard et al, 2007, Tirosh et al, 2007) to CHD risk, which may be particularly important in Latino populations.

The study drug (LOVAZA) improves the TC/HDL ratio which is the strongest predictor of CHD events based on the ~30,000 patient Interheart study noted above. LOVAZA has no hepatic P450 effects and for that matter no meaningful clinical adverse effects, making it advantageous for use in a population with multiple co-morbidities who are at risk for drug-drug interactions and have difficulty with medication adherence. Given the high incidence of insulin resistance among DH's predominately Latino CHD population, and strong lipid (Harris et al, 1997; Davidson et al 2007) as well outcome data in CHD (GISSI investigators, 1999) this agent has potential clinical utility in our population.

To date, improved outcomes in non-CHD populations have not been demonstrated prospectively with LOVAZA. Although recent data suggest promising effects on inflammatory makers such as LpPLA2, the impact of LOVAZA on pre-clinical markers of atherosclerosis such as BAR and CIMT have not been well characterized particularly among Latinos. Moreover, changes in inflammatory markers have been limited and more expansive evaluations are currently available. Against this background we assessed whether LOVAZA might improve atherosclerotic risk via improvement in flow mediated dilation of the brachial artery as well as through reduction in a comprehensive inflammatory marker panel.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HTN
* Hispanic or Non-Hispanic White
* Age > 18
* One additional CVD risk factor

  * Age > 55 for males or >65 for females
  * DM
  * Dyslipidemia O TC >220 or O LDL >130 or O on statin therapy
  * Current smoker
  * Chronic kidney disease defined as GFR <60 ml/min/1.72m2
  * BMI > 30 kg/m2
  * Positive microalbuminuria -Able to sign consent form and willing to complete 12-month follow- up period.

Exclusion criteria used for SA3/4 will also apply for Aim 4.3. These include factors rendering assessment of endothelial function unreliable, such as:

* Clinically manifest CVD (including angina, myocardial infarction, surgical or percutaneous coronary revascularization, stroke, cerebrovascular revascularization, peripheral vascular disease, heart failure, or valvular heart disease
* Electrocardiographic evidence of prior myocardial infarction
* Known valvular heart disease of at least moderate severity
* Known left ventricular systolic dysfunction (LVEF < 0.50)
* End-stage renal disease
* History of inflammatory disease or vasculitis (including rheumatoid arthritis, systemic lupus erythematosis, Raynaud phenomenon, or other connective tissue disease/vasculitides)
* Corticosteroid therapy
* Active substance abuse
* Projected life-expectancy <12 months due to comorbid condition
* Plans to move away from the Denver area within 12 months
* Previous trauma or surgery of the brachial artery
* Upper arm circumference exceeding 42 cm.

Additional exclusion criteria for participation in Aim 4.3 include:

* Pregnancy or breast-feeding
* Known sensitivity or allergy to fish
* Known sensitivity or allergy to omega-3 fatty acid supplements
* Taking omega-3 fatty acid supplements in the last 2 weeks- may participate after 2 week washout
* Triglycerides > 500 mg/dL.
* Alanine aminotransferase (ALT) levels above 3x upper limit of normal
* Not a good candidate for participation based on the opinion of the investigators.
* Current therapy with a fibric acid derivative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlin S Long, MD, Principal Investigator — Denver Health Medical Center Chief of Cardiology
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

REFERENCES:
- [Derived] Krantz MJ, Havranek EP, Pereira RI, Beaty B, Mehler PS, Long CS. Effects of omega-3 fatty acids on arterial stiffness in patients with hypertension: a randomized pilot study. J Negat Results Biomed. 2015 Dec 2;14:21. doi: 10.1186/s12952-015-0040-x. PMID 26631058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was discontinued early due to lack of funding and slow enrollment
Groups:
- Placebo: Placebo (Four 1-gram capsules daily)
- Omega 3: omega-3-acid ethyl esters (Four 1-gram capsules daily)
Period: Overall Study
Arm/Group | Placebo | Omega 3
Started | 42 | 34
Completed | 35 | 27
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omega 3 | Total
Number analyzed (Participants) | 35 | 27 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.8) | 62.3 (9.7) | 61.1 (10.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 22 | 51
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 35 | 27 | 62

OUTCOME MEASURES:

1. Secondary Outcome: Change in Lipoprotein-associated Phospholipase A2 (LpPLA2)
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Omega 3
Number analyzed (Participants) | 35 | 27
ng/mL | -6.1 (31.7) | -18.1 (41.1)
Statistical Analysis 1: Comparison: Placebo vs Omega 3; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis

2. Secondary Outcome: Change in hsCRP
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Omega 3
Number analyzed (Participants) | 35 | 27
mg/L | 0.9 (4.4) | -0.9 (3.1)
Statistical Analysis 1: Comparison: Placebo vs Omega 3; Test type: Superiority or Other; p = 0.08, Mixed Models Analysis

3. Primary Outcome: Change in Pulse Wave Velocity in Active vs. Placebo-treated Patients.
Description: We conducted a prospective, randomized; double-blinded study of omega-3 fatty acids among 60 Latino and White hypertensive patients at risk for CVD. Patients received either 4-g omega-3 fatty acids or matched placebo daily. The principal outcome measure was change in brachial-ankle PWV.
  .
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Placebo | Omega 3
Number analyzed (Participants) | 35 | 27
cm/sec | -33 (306) | -97 (182)
Statistical Analysis 1: Comparison: Placebo vs Omega 3; Test type: Superiority or Other; p = 0.36, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Placebo | Omega 3
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/34
Other Adverse Events (participants affected / at risk) | 0/42 | 0/34

LIMITATIONS AND CAVEATS:
The study was discontinued early due to lack of funding and slow enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall furnish copies of any proposed publication or presentation to the Sponsor for review at least thirty (30) days in advance of the submission of such proposed publication or presentation to a journal, editor or other third party. The sponsor shall have thirty (30) days after receipt of said copies, to object to such proposed presentation or proposed publication.